CLINICAL TRIAL: NCT04308746
Title: Evaluating Attitudes Towards Organ Donation
Brief Title: Evaluating Attitudes Towards Organ Donation in the United States on MTurk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSS-1502-P02-07
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Individual Difference
Keywords: Organ Donation; Culture

STUDY DESIGN:
Intervention Model Description: Participants are assigned to 1 out of 2 culture orientation priming tasks (Individualistic or Collectivistic)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualistic (Experimental): Participants write 3 statements to 3 questions relating to his/her differences from his/her immediate community
  Interventions: Behavioral: Online Individualistic Prime (statement writing)
- Collectivistic (Experimental): Participants write 3 statements to 3 questions relating to his/her similarities with his/her immediate community
  Interventions: Behavioral: Online Collectivistic Prime (statement writing)

INTERVENTIONS:
Behavioral: Online Individualistic Prime (statement writing) — Participants write 3 statements each about (1) themselves, (2) why they are not like others, and (3) why it is beneficial to stand out from others
  Arms: Individualistic
Behavioral: Online Collectivistic Prime (statement writing) — Participants think about a social group and write 3 statements each about (1) their social group, (2) why they are like others, and (3) why it is beneficial to blend in with others
  Arms: Collectivistic

SUMMARY:
The study is conducted to investigate the effects of priming different cultural orientations on participants' decisions on whether to donate their organs, in an opt-out donation system scenario where the default is a presumed consent on the part of the individual.

DETAILED DESCRIPTION:
Participants complete a survey where they respond to scales measuring their baseline cultural and power distance orientations, and answer questions on their demographics such as gender, race, employment etc.

24 hours later, participants fill in a 2nd survey where they are instructed to complete 1 out of 2 possible priming tasks. The possible tasks consist of an Individualistic priming condition and a Collectivistic priming condition; both tasks require participants to answer 3 statements each to 3 questions regarding the self or their social group. Participants then indicate their choice on whether to donate their organs (default or opt-out), rate their confidence regarding their choice and complete the same scales measuring their cultural and power distance orientations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 and above
* Lives in the United States of America

Exclusion Criteria:

* Below age 21
* Does not live in the United States of America

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2020-02-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Binary survey item - Decision to Donate Organ | 1 minute
  From a scenario where participants imagine themselves applying for a driver's license in a country where an opt-out organ donation system is enforced, participants are asked to make a binary choice between choosing to donate their organs (default) and choosing not to donate their organs (opt out).
Line scale survey item - Confidence in Decision to Donate Organ | 1 minute
  Participants are asked to mark along a line scale on how confident they feel about their decision to donate their organs. The extreme ends of the line scale are defined as "Not Confident At All" (0) and "Extremely Confident" (100).

SECONDARY OUTCOMES:
Individual levels of individualism & collectivism | 5 minutes
  Individualism and collectivism levels will be measured by Triandis & Gelfand (1998)'s "Culture Orientation Scale". This is a 16-item scale designed to measure: 1) Vertical Collectivism (VC) - seeing the self as a part of a collective and accepting hierarchy and inequality within that collective; 2) Vertical Individualism (VI) - seeing the self as fully autonomous, but recognizing and accepting the existence of inequality; 3) Horizontal Collectivism (HC) - seeing the self as part of a collective but viewing all the members of that collective as equal counterparts; and 4) Horizontal Individualism (HI) - seeing the self as fully autonomous, and believing in equality amongst individuals.
  All items are answered on a 5-point scale, ranging from 1 = strongly disagree & 5 = strongly agree. Each dimension's items are summed up separately to create a VC, VI, HC, and HI score to reflect the level of collectivism and individualism in the sampled group.
Individual levels of power distance | 3 minutes
  Individualism and collectivism levels will be measured by a 5-item scale used by Hanzaee and Dehkordi (2011) to measure Power Distance, defined as "the extent to which the less powerful members of institutions and organizations within a country expect and accept that power is distributed unequally" (Hofstede and Hofstede, 2005)
  All items are answered on a 5-point scale, ranging from 1 = strongly disagree & 5 = strongly agree. All items are summed up to create an average score to reflect the level of power distance orientation in the sampled group.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided